CLINICAL TRIAL: NCT04818814
Title: SCI Pain App Intervention Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Baylor College of Medicine (Other)
Collaborators: The University of Texas Health Science Center, Houston (Other); TIRR Memorial Hermann (Other)
Responsible Party: Principal Investigator, Susan Robinson Whelen, Principal Investigator, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-47556
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Spinal Cord Injuries; Chronic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Meditation (MM) App (Experimental): Participants randomized to the MM condition will be asked to download and use the free Mindfulness Coach app (available for iOS and Android platforms) developed by the Veteran Affairs National Center for PTSD. The app offers written information about mindfulness as well as 12 audio-guided meditations each lasting 8-13 minutes. Participants will attend a live videochat orientation to the study with the research coordinator (RC) to receive assistance in downloading and using the app. Participants will be asked to listen to at least one, and ideally two, audio-guided meditation exercises using the app daily for six weeks. The RC will ask participants to complete weekly logs of their MM app use via a Qualtrics survey sent via email.
  Interventions: Behavioral: Mindfulness Meditation App
- Engagement and Distraction (ED) App (Active Comparator): Participants randomized to the Engagement and Distraction condition will be asked to download and use the free TED Talk app (available for iOS and Android platforms). The app offers many videos of engaging and distracting presentations about technology, entertainment, and design. The research coordinator will work with the participant to create a customized list of Ted Talk videos, each lasting 6-12 minutes, based on participants' personal interests. Participants will be asked to listen to or watch at least one, and ideally two, presentations using the app daily for six weeks. The research coordinator will ask participants to complete weekly logs of their TED Talk app use via a Qualtrics survey sent via email.
  Interventions: Behavioral: Engagement and Distraction App

INTERVENTIONS:
Behavioral: Mindfulness Meditation App — Listening to audio-guided meditation sessions using a mobile app.
  Arms: Mindfulness Meditation (MM) App
Behavioral: Engagement and Distraction App — Listening to engaging and distracting videos of interest to the participant using a mobile app.
  Arms: Engagement and Distraction (ED) App

SUMMARY:
The purpose of this study is to find out if using an app is a feasible and acceptable treatment for chronic pain in persons with spinal cord injury. Participants will have a 50% chance of being asked to listen to 10 minutes of audio-guided meditations using an app each day for six weeks, and a 50% chance of being asked to listen to 10 minutes of engaging and distracting presentations about topics of interest to the individual (TED Talks) for six weeks. All participants will be asked to complete three online surveys about their emotional and physical health lasting 20-30 minutes (one when the participant first enters the study, one six weeks later, and another six weeks later). Additionally, participants will be asked to complete brief (<5 minute) online surveys once a week during the first six weeks of their participation. Participation in this study is very low risk, and participants may not experience any personal benefit from their participation. Participation in this study is entirely voluntary.

ELIGIBILITY:
Inclusion Criteria:

1. are at least 18 years of age
2. have a traumatic SCI of at least 6 months duration
3. have chronic pain [defined as pain lasting at least 3 months with a pain intensity rating of 4 or higher on a 10-point visual analog scale]
4. understand spoken and written English sufficiently to understand the goals, procedures, time involved, and the time involved in participation, participate in the intervention and complete study surveys.

Exclusion Criteria:

1. have a significant visual or hearing impairment that limits their ability to participate in the app/computer-based intervention
2. lack access to and the ability to use a smart phone or smart tablet (e.g., iPad)
3. are unable to provide or obtain an email address for communication
4. practiced any kind of meditation more than once a week in the past 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Feasibility of Daily Practice as assessed by the proportion of assigned home practice completed | Immediately post-intervention (i.e., 6-weeks post-baseline)
  proportion of assigned home practice completed by participants
Feasibility of Immediate Post-Intervention Follow-Up Assessment as assessed by the proportion of participants who complete immediate post-intervention follow up assessment | Immediately post-intervention (i.e., 6-weeks post-baseline)
  proportion of participants who complete immediate post-intervention follow up assessment
Feasibility of 6-Week Follow-Up Assessment as assessed by the proportion of participants who complete 6 weeks post-intervention follow up assessment | 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  proportion of participants who complete 6 weeks post-intervention follow up assessment
Participant Satisfaction as assessed by a satisfaction questionnaire adapted from the Client Satisfaction Questionnaire for Internet-based Interventions (CSQ-I) | Immediately post-intervention (i.e., 6-weeks post-baseline)
  participant reported satisfaction with their assigned condition; scores range from 12-48, with higher scores indicating greater satisfaction

SECONDARY OUTCOMES:
International SCI Pain Basic Data Subset Questionnaire | Immediately post-intervention (i.e., 6-weeks post-baseline) and 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  Self-reported pain intensity and interference on a 0-10 scale with higher scores indicating greater pain intensity and interference
Chronic Pain Acceptance Questionnaire | Immediately post-intervention (i.e., 6-weeks post-baseline) and 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  Self-reported acceptance of pain; scores range from 0-156 with higher scores indicating greater acceptance of pain
Five Facet Mindfulness Questionnaire-Short Form | Immediately post-intervention (i.e., 6-weeks post-baseline) and 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  Self-reported mindfulness; scores range from 24-120 with higher scores indicating greater mindfulness
Patient Health Questionnaire-8 item | Immediately post-intervention (i.e., 6-weeks post-baseline) and 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  Depressive Symptoms; scores range from 0-24 with higher scores indicating greater depression symptoms
Generalized Anxiety Disorder Questionnaire-7 | Immediately post-intervention (i.e., 6-weeks post-baseline) and 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  Anxiety Symptoms; scores range from 0-21 with higher scores indicating greater anxiety symptoms
SCI-QOL Positive Affect and Wellbeing Questionnaire | Immediately post-intervention (i.e., 6-weeks post-baseline) and 6 weeks post-intervention (i.e., 12-weeks post-baseline)
  Self-reported Quality of Life; scores range from 10-50 with higher scores indicating greater quality of life

OTHER OUTCOMES:
Patient Health Questionnaire-2 item | Assessed weekly during the 6-week intervention
  Depressive Symptoms; scores range from 0-6 with higher scores indicating greater depression symptoms
Generalized Anxiety Disorder Questionnaire-2 | Assessed weekly during the 6-week intervention
  Anxiety Symptoms; scores range from 0-6 with higher scores indicating greater anxiety symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- TIRR Memorial Hermann, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IDP available to other researchers, aside from those directly involved in the project (i.e., listed on the study's IRB protocol at Baylor College of Medicine and the collaborating site, The University of Texas Health Science Center at Houston).